CLINICAL TRIAL: NCT04965675
Title: Interventional, Randomized, Double-blind, Parallel-group, Placebo-controlled Study to Evaluate the Efficacy and Safety of IV Eptinezumab in Adolescents (12-17 Years) for the Preventive Treatment of Chronic Migraine
Brief Title: A Study With Eptinezumab in Adolescents (12-17 Years) With Chronic Migraine
Acronym: PROSPECT-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19356A; 2020-001009-22 (EudraCT Number); 2024-510656-13-00 (EU CTIS Number)
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Chronic Migraine in Children
MeSH Terms: interventions — eptinezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Eptinezumab 300 mg (Experimental): Participants will receive a single IV infusion of eptinezumab 300 mg (weight adjusted).
  Interventions: Drug: Eptinezumab
- Eptinezumab 100 mg (Experimental): Participants will receive a single IV infusion of eptinezumab 100 mg (weight adjusted).
  Interventions: Drug: Eptinezumab
- Placebo (Placebo Comparator): Participants will receive a single IV infusion of placebo matching to eptinezumab.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eptinezumab — Eptinezumab will be administered per dose and schedule specified in the arm.
  Other Names: Vyepti
  Arms: Eptinezumab 100 mg; Eptinezumab 300 mg
Drug: Placebo — Placebo matching to eptinezumab will be administered per schedule specified in the arm.
  Arms: Placebo

SUMMARY:
To find out if eptinezumab is better than placebo (normal saline solution) in lowering the number of days with migraine in young people ages 12 to 17 with chronic migraine.

DETAILED DESCRIPTION:
The study includes a single intravenous (IV) infusion of the study drug and consists of a screening period (4 weeks), a double-blind, placebo-controlled period (12 weeks), and a safety follow-up period (8 weeks). Participants confirmed eligible will be randomized (1:1:1) to receive a single IV infusion of either eptinezumab 300 milligrams (mg) dose (weight adjusted; targeting adult exposure after 300 mg IV), eptinezumab 100 mg (weight adjusted; targeting adult exposure after 100 mg IV), or placebo at randomization visit. The doses will be adjusted for the participant's body weight.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a diagnosis of migraine (with or without aura) as defined by International Classification of Headache Disorders 3 (ICHD-3) guidelines with history of chronic migraine, of at least 6 months prior to the screening visit.
* During the 28-day screening period, the participant must adequately complete the headache eDiary on at least 23 of the 28 days following the screening visit.
* During the 28-day screening period, the participant must have ≥15 to ≤26 headache days, of which at least 8 are migraine days as documented in the eDiary.

Exclusion Criteria:

* The participant has previously been randomised in this study and exposed to eptinezumab.
* The participant has been exposed to any monoclonal antibody treatment (including exposure in a study) <6 months prior to the screening visit.
* The participant has been exposed to another calcitonin gene-related peptide (CGRP) antibody (including exposure in a study investigating a CGRP antibody) <6 months prior to the screening visit.
* The participant has a history or diagnosis of complicated migraine (ICHD-3 version, 2018), chronic tension-type headache, hypnic headache, cluster headache, hemicrania continua, new daily persistent headache, or unusual migraine subtypes such as hemiplegic migraine (sporadic and familial), migraine with brainstem aura, ophthalmoplegic migraine, or migraine with neurological accompaniments that are not typical of migraine aura (diplopia, altered consciousness, or long duration; for example >60 minutes).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 285 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2026-09-05 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Monthly Migraine Days (MMDs) Averaged Over Weeks 1-12 | Baseline, Weeks 1-12

SECONDARY OUTCOMES:
Percentage of Participants With 50% Reduction From Baseline in MMDs Averaged Over Weeks 1-12 | Baseline up to Weeks 1-12
Percentage of Participants With Migraine on the Day After Dosing (Day 1) | Day 1
Change From Baseline in MMDs With Use of Acute Medication Averaged Over Weeks 1-12 | Baseline, Weeks 1-12
Percentage of Participants With 75% Reduction From Baseline in MMDs Averaged Over Weeks 1-12 | Baseline up to Weeks 1-12
Percentage of Participants With 75% Reduction From Baseline in MMDs Averaged Over Weeks 1-4 | Baseline up to Weeks 1-4
Percentage of Participants With 50% Reduction From Baseline in MMDs Averaged Over Weeks 1-4 | Baseline up to Weeks 1-4
Change From Baseline in Monthly Headache Days Averaged Over Weeks 1-12 | Baseline, Weeks 1-12
Change From Baseline in Rate of Migraines With Severe Pain Intensity Averaged Over Weeks 1-12 | Baseline, Weeks 1-12
Change From Baseline in Days With Use of Acute Medication Averaged Over Weeks 1-12 | Baseline, Weeks 1-12
Change From Baseline in Pediatric Migraine Disability Assessment Questionnaire (PedMIDAS) Score Averaged Over Weeks 1-12 | Baseline, Weeks 1-12
Free Eptinezumab Plasma Concentration | Randomization ( pre-dose [Week 0]), Week 8, Week 12, and safety follow up visit (Week 20)
Number of Participants With Specific Anti-Eptinezumab Antibodies (Anti-Drug Antibodies [ADA]) | From randomization (Week 0) up to Week 20
Number of Participants With Specific Anti-Eptinezumab Antibodies for Neutralizing Activity (NAb) | From randomization (Week 0) up to Week 20

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (83):
- United States (21):
  - Yale-New Haven Children's Hospital - PIN, New Haven, Connecticut
  - Ki Health Partners LLC DBA New England Institute for Clinical Research, Stamford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - A G A Clinical Trials, Hialeah, Florida
  - Axcess Medical Research, Loxahatchee Groves, Florida
  - University of South Florida, Tampa, Florida
  - University of Kentucky HealthCare (UKHC) Kentucky Clinic, Lexington, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Michigan State University - Department of Neurology, East Lansing, Michigan
  - Corewell Health Butterworth Hospital, Grand Rapids, Michigan
  - Dent Neurosciences Research Center Incorporated, Amherst, New York
  - North Suffolk Neurology-Commack, Commack, New York
  - OnSite Clinical Solutions, LLC - Randolph Rd - Charlotte, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center - PIN, Cincinnati, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Road Runner Research Ltd, San Antonio, Texas
  - Children's Specialty Group, Norfolk, Virginia
  - Mary Bridge Children's Hospital - PIN, Tacoma, Washington
  - Marshall University Medical Center, Huntington, West Virginia
- Argentina (10):
  - Hospital Privado de La Comunidad, Mar del Plata, Buenos Aires
  - Clínica Privada Independencia, Munro, Buenos Aires
  - Expertia S.A- Mautalén Salud e Investigación, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Hospital Britanico de Buenos Aires, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Hospital Italiano de Buenos Aires, Ciudad Autónoma Buenos Aires, Ciudad Autónoma de BuenosAires
  - Sanatorio Allende S.A, Córdoba, Córdoba Province
  - Hospital de Niños de La Santisima Trinidad, Córdoba-Barrio Crisol, Córdoba Province
  - Instituto Médico Río Cuarto, Río Cuarto, Córdoba Province
  - INECO Neurociencias Oroño, Rosario, Santa Fe Province
  - Centro de Investigaciones Médicas Tucumán - PPDS, San Miguel de Tucumán, Tucumán Province
- Canada (5):
  - University of Alberta, Edmonton, Alberta
  - Medical Arts Health Research Group - Penticton, Penticton, British Columbia
  - Vancouver Island Health Authority, Victoria, British Columbia
  - The Kids Clinic, Ajax, Ontario
  - London Health Sciences Centre -800 Commissioners Rd E, London, Ontario
- Italy (8):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico, Bari, Apulia
  - Ospedale Pediatrico Bambino Gesù IRCCS, Rome, Lazio
  - IRCCS Istituto Giannina Gaslini, Genoa, Liguria
  - Ospedale San Raffaele S.r.l. - INCIPIT - PIN, Milan, Lombardy
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Lombardy
  - Fondazione Istituto Neurologico Nazionale Casimiro Mondino IRCCS, Pavia, Lombardy
  - AO Brotzu - Clinica di Neuropsichiatria dell'Infanzia e dell'Adolescenza - INCIPIT - PIN, Cagliari, Sardinia
  - Azienda Ospedaliero Universitaria A Meyer - INCIPIT - PIN, Florence, Tuscany
- Mexico (9):
  - Centro de Investigacion Medico Biologica y de Terapia Avanzada S.C., Guadalajara, Jalisco
  - Unidad de Investigación en Salud de Chihuahua S.C., Zapopan, Jalisco
  - Centro de Investigacion Clinica Chapultepec S.A. de C.V. - Morelia, Morelia, Michoacán
  - ICARO Investigaciones en Medicina, S.A de C.V, Chihuahua City
  - Neurociencias Estudios Clinicos S.C., Culiacán Sinaloa
  - Instituto de Investigationes Clinicas para la Salud A.C., Durango
  - Unidad de Investigación en Salud de Chihuahua S.C.-Mexico city, Mexico City
  - Clinical Research Institute SC-Mexico, Tepetlacolco
  - Centro de Estudios Clinicos Y Especialidades Medicas SC, Vista Hermosa
- Poland (7):
  - AthleticoMed, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - ETG Neuroscience - PPDS, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Plejady Magdalena Celinska - Lowenhoff, Michal Zolnowski Spolka komandytowa, Krakow
  - ETG Lublin - PPDS, Lublin
  - Instytut Zdrowia Dr Boczarska-Jedynak Sp. z o.o. Sp. k., Oświęcim
  - MTZ Clinical Research Powered by PRATIA - PPDS, Warsaw
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak, Wroclaw
- Portugal (3):
  - ULS de Almada-Seixal, EPE - Hospital Garcia de Orta, Almada, Setúbal District
  - ULS de Coimbra, EPE - Hospital Pediátrico de Coimbra, Coimbra
  - ULS de São João, EPE - Hospital de São João, Porto
- Serbia (4):
  - Childrens University Hospital, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - Children and Youth Health Care Institute of Vojvodina, Novi Sad
  - Clinical Centre of Vojvodina, Novi Sad
- Spain (6):
  - CHUVI - H.U. Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Instituto del Sueño, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Turkey (Türkiye) (5):
  - Izmir City Hospital, Bayraklı, İzmir
  - Eskisehir Osmangazi Universitesi Tip Fakultesi Hastanesi, Eskişehir
  - Istanbul Üniversitesi, Istanbul Tip Fakültesi, Nör, Fatih/Istanbul
  - Istanbul University Cerrahpasa Medical Faculty Hospital, Fatih/Istanbul
  - Mersin University Medical Faculty, Mersin
- United Kingdom (5):
  - Royal Devon and Exeter Hospital NHS Trust - PPDS, Exeter, Devon
  - Queen Elizabeth University Hospital - PPDS, Glasgow, Lanarkshire
  - Great Ormond Street Hospital - PPDS, London, London, City of
  - Royal Hospital for Children and Young People - PIN, Edinburgh, Midlothian
  - James Paget University Hospitals NHS Foundation Trust, Great Yarmouth, Norfolk